CLINICAL TRIAL: NCT00516672
Title: A Phase I, Open-Label, Multiple Dose of Pazopanib Alone and In Combination With Lapatinib in Japanese Patients With Solid Tumors
Brief Title: Phase I Study of Pazopanib Alone and In Combination With Lapatinib in Japanese Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109693
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: lapatinib,; cancer; pharmacokinetics,; safety,; pazopanib,; Japanese patients,
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — pazopanib; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Pazopanib monotherapy or in combination with lapatinib
  Interventions: Drug: pazopanib; Drug: Lapatinib

INTERVENTIONS:
Drug: pazopanib — Pazopanib oral tablet
Drug: Lapatinib — Lapatinib oral tablet

SUMMARY:
This is a two part phase I study in Japanese patients that will determine the safety, tolerability and pharmacokinetics of pazopanib monotherapy and of pazopanib in combination with lapatinib.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent.
* Histologically or cytologically confirmed diagnosis of advanced solid tumor.
* Women and men with potential to have children must be willing to practice acceptable methods of birth control during the study.
* ECOG performance status of 0 or 1.
* Adequate bone marrow reserve and hepato-renal function.
* Able to swallow and retain oral medication.
* For combo part, left ventricular ejection fraction within normal range or above 50%.

Exclusion criteria:

* Prior treatment with pazopanib, and with lapatinib for combo part.
* Clinically significant gastrointestinal abnormalities.
* Sevier diseases or conditions other than cancer.
* Poorly controlled hypertension.
* Use of warfarin for therapeutic anticoagulation.
* Use of other anti-angiogenesis agents, and other ErbB inhibitors for combo part.
* Unresolved and/or unstable toxicities
* Pregnant or lactating females

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09-10 (Actual); Primary Completion 2010-08-30 (Actual); Study Completion 2015-10-14 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | before and after taking the study medications
  The safety and tolerability endpoints will consist of the evaluation of adverse events (AEs), and changes in vital signs and laboratory values.

SECONDARY OUTCOMES:
Pharmacokinetics | over a 24 hour period
  The pharmacokinetic parameters AUC0-24, AUC0-inf (Day 1 only), Cmax, tmax, and t1/2 of pazopanib and its four metabolites. To determine if target trough plasma concentration of pazopanib of 20,000 ng/ml is achieved.
Tumor response | 9 weeks
  Assessments of tumor response will be obtained every 9 weeks and will be recorded as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Saitama

REFERENCES:
- [Derived] Inada-Inoue M, Ando Y, Kawada K, Mitsuma A, Sawaki M, Yokoyama T, Sunakawa Y, Ishida H, Araki K, Yamashita K, Mizuno K, Nagashima F, Takekura A, Nagamatsu K, Sasaki Y. Phase 1 study of pazopanib alone or combined with lapatinib in Japanese patients with solid tumors. Cancer Chemother Pharmacol. 2014 Apr;73(4):673-83. doi: 10.1007/s00280-014-2374-3. Epub 2014 Jan 24. PMID 24464355
- See also: Results for study 109693 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/109693?search=study&search_terms=109693#rs